CLINICAL TRIAL: NCT07385950
Title: Evaluation of Diagnostic Efficacy of a αvβ6/FAP-Targeting Heterodimeric Probe in Patients With Malignant Solid Tumors: An Open-Label, Single-Arm, Single-Center Study
Brief Title: Evaluation of the Diagnostic Efficacy of a αvβ6/FAP-Targeting Heterodimeric Probe in Patients With Malignant Solid Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Yong He, Department of Nuclear Medicine, Zhongnan Hospital of Wuhan University, Zhongnan Hospital
Other Study IDs: IIT2025383
Record Dates: First submitted 2026-01-05; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: PET / CT; Solid Tumors; Adult
Keywords: integrin αVβ6; FAP; PET imaging; Diagnostic efficacy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Recipients with Malignant solid tumors: Participants:
  Patients (≥18 years) with highly suspected or pathologically confirmed malignant tumors, or patients with suspected recurrence of malignant tumors after treatment
  Interventions:
  68Ga-B6FA-01 PET/CT scan prior to therapy.
  Objectives:
  * Evaluate the diagnostic efficacy of 68Ga-B6FA-01 PET in malignant solid tumors.
  * Evaluate the safety and tolerability, biological distribution, radiation dose, and pharmacokinetic characteristics of 68Ga-B6FA-01 in cancer patients.
  * Evaluate the relationship between quantitative parameters of PET imaging and pathological indicators Design: Single-arm observational study; PET parameters (SUVmax, tumor-to-background ratio, et al) will be correlated with clinical outcomes.
  Interventions: Diagnostic Test: PET/CT Imaging with αvβ6/FAP-targeted tracer

INTERVENTIONS:
Diagnostic Test: PET/CT Imaging with αvβ6/FAP-targeted tracer — Intravenous administration of αvβ6/FAP-targeted tracer (111~185 MBq), followed by whole-body PET/CT scan 30~60 minutes post-injection.

SUMMARY:
Malignant tumors pose a grave threat to human health and impose a substantial burden on society. Molecular imaging, which enables non-invasive, in vivo visualization of biological processes at the molecular level, is crucial for early diagnosis and treatment monitoring, thereby improving clinical management. Currently, molecular probes targeting fibroblast activation protein (FAP) and integrin αvβ6, such as ⁶⁸Ga-labeled FAPI and ⁶⁸Ga-Trivehexin, have shown promise in oncologic PET imaging, yet each has limitations.

FAP is predominantly overexpressed in cancer-associated fibroblasts within the tumor stroma, with minimal expression in normal tissues. However, radiotracers like ⁶⁸Ga-FAPI often exhibit physiological uptake in normal organs (e.g., salivary glands, pancreas, uterus), leading to elevated background signals and potentially reduced diagnostic contrast. Conversely, integrin αvβ6 is primarily expressed on tumor cell surfaces and is upregulated in many malignancies. Nonetheless, probes like ⁶⁸Ga-Trivehexin suffer from high renal retention with slow clearance and notable physiological gastrointestinal uptake, resulting in suboptimal target-to-background ratios and compromised image quality.

Given the complementary expression profiles of FAP (stroma) and integrin αvβ6 (tumor cells), we hypothesize that a bispecific molecular probe capable of simultaneously engaging both targets could achieve superior tumor targeting through a synergistic "dual-lock" mechanism. This prospective exploratory clinical trial aims to evaluate the diagnostic efficacy and safety of a novel bispecific probe, named ⁶⁸Ga-B6FA-01, in patients with malignant solid tumors. The ultimate goal is to develop a superior imaging strategy for early and precise tumor diagnosis, treatment response assessment, and personalized therapeutic decision-making.

DETAILED DESCRIPTION:
This investigator-initiated trial (IIT) aims to evaluate the clinical utility of positron emission tomography (PET) imaging targeting both integrin αvβ6 and fibroblast activation protein (FAP) in patients with malignant solid tumors. Based on promising preclinical studies, we have designed and synthesized a bispecific probe, B6FA-01, which can simultaneously bind to both targets. By concurrently targeting two independent, highly expressed targets-one on tumor epithelial cells (αvβ6) and one within the tumor stroma (FAP)-this probe is expected to address the issue of receptor heterogeneity that limits current single-target probes like ⁶⁸Ga-FAPI or ⁶⁸Ga-Trivehexin. Indeed, preclinical data indicate that ⁶⁸Ga-B6FA-01 exhibits not only excellent targeting affinity and specificity but also higher tumor uptake, longer intratumoral retention, faster renal clearance, and a favorable biocompatibility profile compared to its single-target counterparts.

In this prospective study, patients with histologically confirmed malignant solid tumors will undergo ⁶⁸Ga-B6FA-01 PET/CT imaging. Key PET parameters-including the maximum standardized uptake value (SUVmax), mean standardized uptake value (SUVmean), and tumor-to-background ratio (TBR)-will be analyzed to assess their diagnostic performance (sensitivity, specificity, accuracy). Furthermore, the study will explore the correlation between these in vivo imaging parameters and the ex vivo expression levels of αvβ6 and FAP in tumor tissues.

The findings from this study could establish αvβ6- and FAP-targeted PET imaging as a superior, non-invasive tool for tumor diagnosis and treatment assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provide written informed consent.
2. Age ≥ 18 years.
3. Newly diagnosed with a clinically/radiologically suspected or pathologically confirmed malignant solid tumor, or with suspected recurrence after prior treatment.
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1.
5. Life expectancy > 6 months.
6. Participants of childbearing potential and their partners must agree to use highly effective contraception for 6 months following the last dose of the investigational agent.

Exclusion Criteria:

1. Prior radioisotope therapy within an interval less than 10 times the physical half-life of the respective radionuclide before study administration.
2. Concurrent participation in any other interventional clinical trial.
3. Known allergy or hypersensitivity to the investigational agent or any of its excipients.
4. Inability to lie still for the duration of the PET scan or any condition contraindicating PET imaging.
5. Pregnancy or lactation.
6. Any other condition that, in the investigator's judgment, would compromise participant safety or study integrity.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants must voluntarily enroll and provide written informed consent, be aged 18 to 90 years (inclusive) regardless of gender, and have a pathologically confirmed diagnosis of treatment-naïve malignant solid tumors or suspected of having a recurrence after treatment. Additionally, participants must demonstrate willingness and ability to comply with scheduled clinical visits.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic sensitivity and specificity of 68Ga-B6FA-01 PET/CT in the staging of malignant tumors | 3 years
  To assess the he diagnostic performance of 68Ga-B6FA-01 PET/CT in patients with newly diagnosed malignancies. Accuracy will be evaluated using a composite reference standard, including histopathological confirmation, clinical follow-up, and additional imaging findings.

SECONDARY OUTCOMES:
The connection between B6FA-01 PET parameters and histopathological biomarkers. | Within 4 weeks of B6FA-01 PET scan
  Analyze the correlation between B6FA-01 PET parameters (SUVmax/SUVmean/SUVpeak, measured in the Syngo Workstation (Siemens Healthineers)) and FAP and αVβ6 expression levels (H-score; immunohistochemistry) or immune - related biomarkers, such as PD-L1 expression (Combined Positive Score; Dako 22C3 IHC assay), CD8 expression (H-score; immunohistochemistry).

CONTACTS AND LOCATIONS:
Overall Officials: Yong He, MD, PhD, Principal Investigator — Zhongnan Hospital
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
The data sharing plan for individual participant data (IPD) from this single-center, investigator-initiated trial has not yet been finalized. The decision will depend on several factors, including the final data governance policies of Zhongnan Hospital of Wuhan University, future intellectual property considerations, and the specific requirements of potential collaborative or publication opportunities. A formal plan will be developed in accordance with institutional guidelines and prevailing best practices for data sharing in clinical research. Data may potentially be made available upon reasonable request and subject to appropriate ethical and administrative approvals.

REFERENCES:
- [Background] Zang J, Wen X, Lin R, Zeng X, Wang C, Shi M, Zeng X, Zhang J, Wu X, Zhang X, Miao W, Xu P, Guo Z, Zhang J, Chen X. Synthesis, preclinical evaluation and radiation dosimetry of a dual targeting PET tracer [68Ga]Ga-FAPI-RGD. Theranostics. 2022 Oct 9;12(16):7180-7190. doi: 10.7150/thno.79144. eCollection 2022. PMID 36276644